CLINICAL TRIAL: NCT06815588
Title: Improving the Outcomes of Children With Tuberculosis Through Innovative Diagnostics and Treatment Monitoring
Acronym: RoGer Pedi
Status: Recruiting | Type: Observational
Sponsor: Research Center Borstel (Other)
Collaborators: LMU Klinikum (Other)
Responsible Party: Sponsor
Other Study IDs: EESS - RoGer Pedi
Record Dates: First submitted 2024-12-17; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-01

CONDITIONS: Tuberculosis
Keywords: pediatric TB; non-sputum diagnosis; post TB lung disease
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Biospecimen Retention: Samples With DNA — Stool samples, mask samples (exhaled air), blood (for biomarkers only)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study aims at identifying and evaluating novel diagnostic methods for children evaluated for respiratory tuberculosis. The investigators will use alternative samples like stool, urine, and masks to diagnose children with respiratory tuberculosis. Once diagnosed, the investigators will use target next generation sequencing to determine if the bacillus is resistant to any of the drugs used for treatment. Additionally, children initiated under TB treatment will be followed-up during treatment to measure blood biomarkers for outcome prediction. Finally, spirometry will be performed longitudinally until 3 months after the end of treatment to assess the lung capacity of children treated for respiratory TB. All children initiated on TB treatment will fill in a quality of life questionnaire.

DETAILED DESCRIPTION:
Tuberculosis (TB) remains a significant global health concern, particularly among children, who are especially vulnerable, with an estimated 1.25 million incident cases and 214,000 deaths reported in 2022. TB in children presents unique challenges due to its subtle clinical manifestations and paucibacillary nature, often resulting in difficulties in diagnosis. Compared to estimated incidence, only 49% children were diagnosed and reported, with the highest proportion of under-reporting taking place in children under 5 years - of 58%. Gaps and challenges persist in accurately diagnosing and treating TB in children, stemming from limitations in traditional diagnostic methods, like sputum culture, that often lack sensitivity and specificity in children. Therefore, there is a pressing need to identify new diagnostic techniques that are both accurate and feasible in pediatric settings.

In recent years, researchers have explored innovative approaches, including the utilization of alternative sample types such as mask samples, urine, or stool, for TB diagnosis in children. These alternative samples offer potential advantages in terms of ease of collection and potentially improved diagnostic accuracy. In 2021, the World Health Organization (WHO) recommended stool as an alternative sample for TB diagnosis in children with signs and symptoms of TB, since stool is non-invasive and easy to collect even in young children. A recent systematic review showed that Xpert Ultra summary sensitivity verified by culture was 56.1% (95% CI 39.1 to 71.7), and specificity was 98.0% (95% CI 93.3 to 99.4), nevertheless the sensitivity results are highlighted as "moderate quality evidence", therefore more research is needed on the performance of this alternative sample in children for the diagnosis of tuberculosis. Moreover, the lipoarabinomannan (LAM) found in the membrane of the Mycobacterium tuberculosis bacillus can be identified in urine and pilot data generated by our group shows a sensitivity of 66% in adults with culture-confirmed pulmonary tuberculosis. This urine-based assay can be critically useful in the diagnosis of extrapulmonary TB as it's not sputum-based. In addition to stool and urine, another promising sample can be obtained through a gelatin strip inside a mask worn by children with presumptive TB. The exhaled breath potentially containing M. tuberculosis bacilli is then captured on the gelatin filter, processed, and tested using GeneXpert.

Once the tuberculosis diagnosis is made, an important challenge lies in drug susceptibility testing (DST), in case of multi-drug resistant TB or rifampicin-resistant TB (MDR/RR-TB)(6). The standard of care for DST is sputum culture, which has many challenges in children, as highlighted above. Targeted next-generation sequencing (tNGS) has emerged as a promising tool for assessing drug sensitivity, providing valuable insights into personalized treatment regimens for pediatric TB cases. In addition, tNGS can be performed on clinical samples like sputum or stool with the potential of a rapidly-available result informing the choice of regimen and clinical decision-making.

After treatment initiation, a main concern lies in treatment monitoring, this step being especially challenging in children. Transcriptomics holds promise for monitoring treatment response in children with TB. By examining gene expression patterns, transcriptomic analyses can offer valuable insights into the efficacy of treatment regimens and help identify early indicators of treatment failure or relapse. Both WHO definitions and TBnet definitions will be used to assess TB outcomes.

Understanding and assessing the burden of post-TB sequelae in children is crucial for ensuring comprehensive care and addressing long-term health outcomes. Therefore, studying and evaluating port-TB disease in children is imperative for improving clinical management strategies and enhancing the overall health outcomes of pediatric TB patients. Spirometry will be used to assess pulmonary function in children.

This study aims to research a novel and comprehensive approach to TB diagnosis, treatment adaptation, and treatment monitoring in the pediatric population, with the overall goal of improving TB outcomes in children.

Aims and objectives

Aim: Improve the diagnosis of tuberculosis and treatment outcomes in children evaluated for tuberculosis

Specific objectives:

1. Identify the diagnostic accuracy of mask strip samples against a composite reference standard for the diagnosis of respiratory tuberculosis in children.
2. Determine the diagnostic accuracy of a novel urinary LAM assay against a composite reference standard for the diagnosis of respiratory tuberculosis in children.
3. Evaluate the diagnostic accuracy of stool and perform targeted next generation sequencing from stool for drug sensitivity testing.
4. Assess the utility of a transcriptomic signature for treatment monitoring and treatment shortening in children treated for respiratory tuberculosis.
5. Measure the pulmonary function changes in children diagnosed with respiratory tuberculosis using spirometry.
6. Assess the quality of life of children treated for respiratory tuberculosis at baseline, during, and after treatment.

ELIGIBILITY:
Inclusion criteria

* Children under 15 years evaluated for respiratory TB.
* Signature of the informed consent form by the parent/guardian and assent form by the child if applicable.

Exclusion criteria

- Refusal to sign informed consent

Ages: 0 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: All potential participants presenting with the inclusion criteria, will be asked to participate in the study upon their parent/guardian consent and their assent, if applicable. Information will be provided about the study and the risks and benefits of participating. Both the child and the parent/guardian are then asked to consent (or assent) to the participation in the study and any questions they might have are answered. The enrollment is complete after the signature of the informed consent form (ICF). If the child or their parent/guardian does not wish to participate in the study, they will receive the standard of care.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-09-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Stool diagnostic accuracy | at baseline
  Evaluate the diagnostic accuracy of stool and perform targeted next generation sequencing from stool for drug sensitivity testing.

SECONDARY OUTCOMES:
Biomarkers for treatment monitoring | from baseline to 9 months pos-enrollment (6 months of treatment + 3 months follow-up post-treatment)
  Assess the utility of a transcriptomic signature composed of a 22-gene RNA model (TB22 - PMID: 33574078) for treatment monitoring and treatment shortening in children treated for respiratory tuberculosis.
Masks diagnostic accuracy | baseline
  Identify the diagnostic accuracy of mask strip samples against a composite reference standard for the diagnosis of respiratory tuberculosis in children.
Urinary LAM diagnostic accuracy | baseline
  Determine the diagnostic accuracy of a novel urinary LAM assay against a composite reference standard for the diagnosis of respiratory tuberculosis in children.
Post-TB lung disease assessment | from baseline to 9 months post-enrollment (6 months of treatment + 3 months follow-up post-treatment)
  Measure the forced vital capacity as a marker of lung function in children diagnosed with respiratory tuberculosis using spirometry.
Quality of life assessment | from baseline to 9 months post-enrollment (6 months of treatment + 3 months follow-up post-treatment)
  Assess the quality of life of children treated for respiratory tuberculosis at baseline, during, and after treatment, using the validated PedsQL questionnaire translated into Romanian and adapted to each age (only the parents respond to the questionnaire for 1-12 months, or 13-24 months; both children and parents respond to the questionnaire for 2-4, or 5-7, or 8-12, or 13-15 years). Higher scores translate to a poorer quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Lange, Professor, Principal Investigator — Research Center Borstel
Locations (1):
- Marius Nasta Institute of Pneumology, Bucharest, BUC, Romania

IPD SHARING:
Plan to Share IPD: Yes
IPD can be shared upon specific request from the study sponsor and after a written agreement is signed
Supporting Information: Study Protocol, ICF
Time Frame: from 2024 to 2034
Access Criteria: anyone contacting the study sponsor, upon written signature of a data sharing agreement